CLINICAL TRIAL: NCT06666842
Title: Longitudinal Effects of a Digital WM Program on Weight Loss: a Randomized Controlled Trial
Brief Title: Longitudinal Effects of a Commercial Digital Weight Management Program on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noom Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00064357
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Weight Loss; Weight Maintenance; Digital Health; Mobile App
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two conditions in a parallel design with assessments occurring before randomization (Baseline) and at 16, 29, 42, and 68 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Noom Weight (Experimental): Participate in a 16-week fully remote digital weight management program focusing on weight loss and management via behavioral change
  Interventions: Behavioral: Noom Weight
- Educational Control (Active Comparator): Receive 16 weekly weight loss-related educational emails based on the United States Department of Agriculture (USDA) Dietary Guidelines
  Interventions: Behavioral: Educational Control

INTERVENTIONS:
Behavioral: Noom Weight — Participants assigned to Noom Weight will be provided access to the app-based program for 16 weeks. This program offers access to self-monitoring features, psychoeducational articles, one-on-one coaching from health experts, and group support. The app includes a robust database of foods, allowing users to track their energy intake. Self-monitoring via the app enables users to review and monitor behavior and weight change patterns. Daily articles review principles of behavior change, nutrition, exercise, etc.
  Arms: Noom Weight
Behavioral: Educational Control — Participants assigned to the educational control will receive 16 brief (5-10 minute read) weekly newsletters outlining information on developing and maintaining a healthy diet and lifestyle adapted from the 2015-2020 Department of Health and Human Services (HHS) and Department of Agriculture (USDA) Dietary Guidelines for Americans. Newsletters include detailed information on topics such as nutrition fundamentals (e.g., calorie limits; healthy eating), food groups and dietary guidelines (e.g., importance of vegetables, fruits, and grains), and tips for habit change (e.g., reducing added sugar and saturated fats). Each week includes prompts for individuals to try new strategies (e.g., make a conscious decision about everything you eat; try to eat at your calorie budget).
  Arms: Educational Control

SUMMARY:
This randomized controlled trial (RCT) will test how well a fully remote weight management program (Noom Weight) helps adults with overweight or obesity (BMI 25-45) achieve weight loss in both the short-term (16 weeks) and the long-term (68 weeks), compared to an educational program). Participants will be randomly assigned to use the 16-week Noom Weight program or receive weekly emails with weight loss-related tips and information. Weight will be measured at baseline, 16, 29, 42, and 68 weeks. Changes in physical activity, eating disorder risk, and body appreciation will also be assessed.

DETAILED DESCRIPTION:
The proposed study seeks to rigorously evaluate and compare the effectiveness of a fully remote digital weight management program (Noom Weight) to an educational control.

Potential participants will be recruited via social media advertisements, which include a brief study description, eligibility criteria, and a link to a web-based screening questionnaire to assess eligibility and interest. If deemed eligible, participants will be invited to complete informed consent and baseline questionnaires. Study staff will then use a random number generator to allocate participants randomly to the Noom Weight program or the educational control. All participants will receive a cellular-connected digital scale (Body Trace), which will be linked to participant IDs and synced to record weigh-ins automatically.

During the initial 16 weeks, Noom Weight participants will be invited to engage with the mobile-based app, which focuses on weight loss and management via behavioral change, and provides features such as self-monitoring, psychoeducational articles, one-on-one coaching from health experts, and group support. Educational control participants will receive 16 weekly weight loss-related educational emails based on the United States Department of Agriculture (USDA) Dietary Guidelines.

After completing the program at 16 weeks, participants will be asked to complete an online questionnaire assessing weight, physical activity, eating disorder risk, and body appreciation. Additional data collection will occur via online questionnaires at 29, 42, and 68 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old
* Self-reported body mass index (BMI) of 25-45
* Proficient in English
* Live in the United States
* Have access to an iOS smartphone or tablet and were willing to use applications daily
* Willing to abstain from engaging in other weight loss programs for 16 weeks
* Willing to discontinue any current over-the-counter (OTC) supplements not recommended/prescribed by a physician (except for multivitamins or other vitamin supplements)
* Have a goal of losing weight
* Complete a decisional balance exercise based on the work of Goldberg and Kiernan (2005). During this exercise, participants reviewed the nature, design, and importance of this study and were prompted to consider the pros and cons of participation. The purpose of this exercise was to ensure that participants fully understood and were willing to participate in the study, as well as to increase study retention.

Exclusion Criteria:

* Weight loss of ≥ 5 kg within the past 6 months
* History of heart problems (e.g., angina, bypass surgery, myocardial infarction, etc.) within the past 6 months
* Major surgery interfering with consuming a regular diet and performing physical activity within the past 6 months
* Hospitalized for psychiatric problems within the past 12 months
* Paid subscription to Noom within the past 12 months
* Concurrent enrollment in other weight management programs or clinical trials that may interfere
* Living with another study participant
* Ever been diagnosed with an eating disorder
* Diagnosis of conditions indicative of weight loss difficulties or unsupervised exercise as being unsafe or unreasonable (e.g., orthopedic limitations, heart problems)
* History of chronic/inflammatory gastrointestinal disorder, with the expectation of irritable bowel syndrome
* Diagnosis of diabetes
* Previous surgical procedure for weight loss
* Presence of implanted cardiac defibrillator or pacemaker
* Current, recent, or planned pregnancy in the next 12 months
* Cancer within past 5 years
* Current cancer treatment
* Untreated thyroid disease or changes (type or dose) in thyroid medication in the last 6 months
* Prescription medication with known effects on appetite or weight (e.g., oral steroids, weight loss medications such as Qsymia, Contrave, etc.) with the exception of a stable dose of selective serotonin reuptake inhibitors (SSRIs) for 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Percent weight change at Week 16 | Baseline, Week 16
  Body weight will be measured using self-report and cellular-connected digital scales (Body Trace). The digital scale is linked to participant IDs and synced to record weigh-ins automatically. If a participant does not report a weight or the reported weight appears to be erroneous, then the raw scale data will be used.

SECONDARY OUTCOMES:
Percent weight change at Week 29 | Baseline, Week 29
  Body weight will be measured using self-report and cellular-connected digital scales (Body Trace). The digital scale is linked to participant IDs and synced to record weigh-ins automatically. If a participant does not report a weight or the reported weight appears to be erroneous, then the raw scale data will be used.
Percent weight change at Week 42 | Baseline, Week 42
  Body weight will be measured using self-report and cellular-connected digital scales (Body Trace). The digital scale is linked to participant IDs and synced to record weigh-ins automatically. If a participant does not report a weight or the reported weight appears to be erroneous, then the raw scale data will be used.
Percent weight change at Week 68 | Baseline, Week 68
  Body weight will be measured using self-report and cellular-connected digital scales (Body Trace). The digital scale is linked to participant IDs and synced to record weigh-ins automatically. If a participant does not report a weight or the reported weight appears to be erroneous, then the raw scale data will be used.
Physical activity change at Week 68 | Baseline, Week 68
  Physical activity will be measured by the 7-item short International Physical Activity Questionnaire (IPAQ), which evaluates minutes of walking, moderate-intensity activities, and vigorous-intensity activities in the last seven days. Higher scores indicate more minutes engaging in each category.
Changes in eating disorder risk at Week 68 | Baseline, Week 68
  Eating disorder risk will be measured by the 28-item Eating Disorder Risk Questionnaire (EDE-Q), which evaluates the range, frequency, and severity of behaviors associated with a diagnosis of an eating disorder in the last four weeks using a seven-point Likert scale (1 = No Days; 2 = 1-5 Days; 3 = 6-12 Days; 4 = 13-15 Days; 5 = 16-22 Days; 6 = 23-27 Days; 7 = Every Day). Higher scores indicate greater eating disorder risk, with a global score of 4 or higher indicating a high risk of a clinical eating disorder.
Changes in body appreciation at Week 68 | Baseline, Week 68
  Body appreciation will be measured by the 10-item Body Appreciation Scale-2 (BAS), which evaluates acceptance, respect, and positive attitudes toward one's body using a five-point Likert scale (1 = Never; 2 = Seldom; 3 = Sometimes; 4 = Often; 5 = Always). Higher scores indicate greater body appreciation.

CONTACTS AND LOCATIONS:
Locations (1):
- Noom Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No